CLINICAL TRIAL: NCT03737006
Title: Coxsackievirus Group B (CVB) Infection in Early Pregnancy
Brief Title: Coxsackie Virus in Pregnancy and Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201602122
Record Dates: First submitted 2017-04-11; First posted 2018-11-09 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Congenital Heart Disease in Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1-(HLHS) effected pregnancies: Consent,blood draw, nose swab, stool collection,questionnaire and review of medical records.
- 2-Other Congenital Heart Defect (OCHD): Consent, blood draw, nose swab, stool collection, questionnaire and review of medical records.
- 3-Healthy Controls (UC): Consent, blood draw, nose swab, stool collection, questionnaire and review of medical records.

SUMMARY:
Investigators would like to find out if a woman's exposure to Coxsackievirus has an effect or increase in incidence of babies being born with congenital heart disease(CHD)

DETAILED DESCRIPTION:
The investigator proposes that Coxsackievirus group B (CVB) infection in early pregnancy induces pathological changes in congenital heart defects. To test the hypothesis, it will be determined if the incidence of CVB infection in women with babies that are congenital heart defect-(CHD) affected pregnancies are higher than in control subjects.

After informed consent participants will provide the following samples during one study visit: 10 mL (about 2 teaspoons) blood draw, a nose swab, provide a stool specimen (or have a rectal swab) and complete a study questionnaire Our 3 study groups are the following-Group 1 is Hypoplastic Left Heart Syndrome or HLHS effected pregnancies. Group 2 is OCHD- Other Congenital Heart Defects and Group 3 is Unaffected Controls (UC) also known as healthy controls.

After informed consent participants will provide the following samples: 10 mL (about 2 teaspoons) blood draw, a nose swab, provide a stool specimen (or have a rectal swab).

A health history review and questionnaire will also be obtained.

Analysis of these samples(blood, stool and nose secretions), a medical history review and questionnaire data will help to determine if there is a link or increased risk of those who may be exposed to virus.

Note- Prior to April 2016- the protocol and the healthy control (HC)subjects group were enrolled to come in for three study visits at varying times in their pregnancy. Blood, nose and stool samples were obtained at all three visits.

ELIGIBILITY:
Inclusion Criteria

* Fetal echocardiogram demonstrating one of the following: Hypoplastic Left Heart Syndrome (HLHS) or variant, other congenital heart disease (OCHD), or unaffected control (UC)
* Gestation is ≥20 wks-fetal group (HLHS, OCHD)
* Subject is able and willing to give informed consent.

Exclusion Criteria

* Subject is < 18 years of age.
* Subject is pregnant with twins or multiple gestations.
* Subject's pregnancy is affected by 3 or more congenital anomalies (in addition to the heart defect).
* Subject's pregnancy is affected by chromosomal anomalies (OCHD & UC groups)
* Maternal history of chromosomal anomaly (OCHD & UC groups)
* Infertility treatment for current/index pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Women
Study Population: Pregnant Woman whose babies have been diagnosed with CHD ( a congenital heart defect) and controls (pregnant women babies without CHD).
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Maternal prenatal and newborn Cox B viral strand identification | 3 - 5years
  Virus identification: Comparison to VP1 sequences available in GenBank will be used to identify the strain of CVB in the isolates.
Maternal prenatal and newborn Cox B antibody levels | 3 - 5years
  Serum CVB antibody titers: Past or current CVB infection will be determined from titers (>/= 1:80) collected from stool, serum and a nasal swab.

SECONDARY OUTCOMES:
Variables and trends influencing Congenital Heart Disease | 3-5 years
  Questionnaires and medical records: To account for potential confounders of CVB serology results through exploratory regression type analysis. Preliminary data is needed to investigate the relationship between variables and measured endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Pirooz Eghtesady, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St Louis Childrens Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tchervenkov CI, Jacobs JP, Weinberg PM, Aiello VD, Beland MJ, Colan SD, Elliott MJ, Franklin RC, Gaynor JW, Krogmann ON, Kurosawa H, Maruszewski B, Stellin G. The nomenclature, definition and classification of hypoplastic left heart syndrome. Cardiol Young. 2006 Aug;16(4):339-68. doi: 10.1017/S1047951106000291. PMID 16839428
- [Background] Hickey EJ, Caldarone CA, McCrindle BW. Left ventricular hypoplasia: a spectrum of disease involving the left ventricular outflow tract, aortic valve, and aorta. J Am Coll Cardiol. 2012 Jan 3;59(1 Suppl):S43-54. doi: 10.1016/j.jacc.2011.04.046. PMID 22192721
- [Background] Kallewaard NL, Zhang L, Chen JW, Guttenberg M, Sanchez MD, Bergelson JM. Tissue-specific deletion of the coxsackievirus and adenovirus receptor protects mice from virus-induced pancreatitis and myocarditis. Cell Host Microbe. 2009 Jul 23;6(1):91-8. doi: 10.1016/j.chom.2009.05.018. PMID 19616768
- [Background] Shi Y, Chen C, Lisewski U, Wrackmeyer U, Radke M, Westermann D, Sauter M, Tschope C, Poller W, Klingel K, Gotthardt M. Cardiac deletion of the Coxsackievirus-adenovirus receptor abolishes Coxsackievirus B3 infection and prevents myocarditis in vivo. J Am Coll Cardiol. 2009 Apr 7;53(14):1219-26. doi: 10.1016/j.jacc.2008.10.064. PMID 19341864
- [Background] Bergelson JM, Cunningham JA, Droguett G, Kurt-Jones EA, Krithivas A, Hong JS, Horwitz MS, Crowell RL, Finberg RW. Isolation of a common receptor for Coxsackie B viruses and adenoviruses 2 and 5. Science. 1997 Feb 28;275(5304):1320-3. doi: 10.1126/science.275.5304.1320. PMID 9036860
- [Background] McBride KL, Marengo L, Canfield M, Langlois P, Fixler D, Belmont JW. Epidemiology of noncomplex left ventricular outflow tract obstruction malformations (aortic valve stenosis, coarctation of the aorta, hypoplastic left heart syndrome) in Texas, 1999-2001. Birth Defects Res A Clin Mol Teratol. 2005 Aug;73(8):555-61. doi: 10.1002/bdra.20169. PMID 16007587
- [Background] Delorme-Axford E, Donker RB, Mouillet JF, Chu T, Bayer A, Ouyang Y, Wang T, Stolz DB, Sarkar SN, Morelli AE, Sadovsky Y, Coyne CB. Human placental trophoblasts confer viral resistance to recipient cells. Proc Natl Acad Sci U S A. 2013 Jul 16;110(29):12048-53. doi: 10.1073/pnas.1304718110. Epub 2013 Jul 1. PMID 23818581